CLINICAL TRIAL: NCT05645692
Title: A Phase II, Randomized, Multicenter, Open-Label, Controlled Study of Tobemstomig Alone or in Combination With Tiragolumab Versus Atezolizumab in Patients With Previously Untreated Locally Advanced or Metastatic Urothelial Cancer Who Are Ineligible for Platinum-Containing Chemotherapy
Brief Title: A Study Evaluating Different Immunotherapies (LAG-3 and PD-1 With or Without TIGIT, Compared to PD-L1 Alone) in Participants With Untreated Locally Advanced Metastatic Urothelial Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO44157
Record Dates: First submitted 2022-11-28; First posted 2022-12-09 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Urothelial Cancer
MeSH Terms: interventions — atezolizumab; Tiragolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Active Comparator): Participants will receive intravenous (IV) atezolizumab every 3 weeks (Q3W).
  Interventions: Drug: Atezolizumab
- Arm B (Experimental): Participants will receive IV tobemstomig Q3W.
  Interventions: Drug: Tobemstomig
- Arm C (Experimental): Participants will receive IV tobemstomig + IV tiragolumab Q3W.
  Interventions: Drug: Tobemstomig; Drug: Tiragolumab

INTERVENTIONS:
Drug: Atezolizumab — Participants will receive 1200 mg IV atezolizumab Q3W.
  Arms: Arm A
Drug: Tobemstomig — Participants will receive 600 mg IV tobemstomig Q3W.
  Other Names: RO7247669
  Arms: Arm B; Arm C
Drug: Tiragolumab — Participants will receive 600 mg IV tiragolumab Q3W.
  Arms: Arm C

SUMMARY:
This study will evaluate the safety of tobemstomig alone or in combination with tiragolumab compared with atezolizumab in participants with previously untreated, locally advanced or metastatic urothelial cancer (mUC) who are ineligible to receive a platinum containing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2
* Histologically or cytologically documented locally advanced or metastatic transitional cell carcinoma (TCC) of the urothelium. Participants with squamous, sarcomatoid, micropapillary, and glandular variant histologies are eligible for inclusion in the study, provided that a urothelial component is present in the tumor specimen. Participants with other variant histologies or pure variant histologies are not eligible for inclusion in this study
* Ineligible ("unfit") to receive platinum-based chemotherapy
* No prior chemotherapy for inoperable locally advanced or metastatic or recurrent urothelial carcinoma (UC)
* Measurable disease; at least one measurable lesion as defined by response evaluation criteria in solid tumors, version 1.1 (RECIST v1.1)
* Availability of a representative leftover tumor specimen that is suitable for determination of PD-L1 status as assessed by a central laboratory
* Adequate hematologic and end organ function
* Negative for hepatitis B and hepatitis C virus (HCV)
* Adequate cardiovascular function

Exclusion Criteria:

* Pregnancy or breastfeeding
* GFR <15 mL/min/1.73 m2
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
* History of leptomeningeal disease
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
* Uncontrolled or symptomatic hypercalcemia
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Active tuberculosis (TB) or acute Epstein-Barr virus (EBV)
* Significant cardiovascular/cerebrovascular disease within 3 months prior to initiation of study treatment
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* History of another primary malignancy other than urothelial carcinoma within 2 years prior to initiation of study treatment, with the exception of malignancies with a negligible risk of metastasis or death
* Severe infection within 4 weeks prior to initiation of study treatment
* Treatment with therapeutic oral or intravenous antibiotics within 2 weeks prior to initiation of study treatment. Participants receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease [COPD] exacerbation), or who are receiving oral antibiotics to treat a urinary tract infection are eligible for the study
* Prior allogeneic stem cell or solid organ transplantation
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during treatment or within 5 months after the final dose of atezolizumab, 4 months after the final dose of tobemstomig, or 90 days after the final dose of tiragolumab
* Current treatment with anti-viral therapy for HBV
* Treatment with any approved anti-cancer therapy, including chemotherapy or hormonal therapy, within 3 weeks prior to initiation of study treatment
* Treatment with investigational therapy within 4 weeks or 5 drug-elimination half-lives (whichever is longer) prior to initiation of study treatment
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-TIGIT and anti-LAG3 therapeutic antibodies or pathways targeting agents
* Treatment with systemic immunostimulatory agents within 4 weeks or 5 drug-elimination half-lives prior to initiation of study treatment
* Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse Events | Up to approximately 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-LaRoche
Locations (56):
- United States (2):
  - Cleveland Clinic, Cleveland, Ohio
  - MD Anderson Cancer Center, Houston, Texas
- Australia (3):
  - Macquarie University Hospital, Macquarie Park, New South Wales
  - Lyell McEwin Hospital, Adelaide, South Australia
  - ICON Cancer Care Adelaide, Kurralta Park, South Australia
- Brazil (5):
  - Hospital Universitario Evangelico De Curitiba, Curitiba, Paraná
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital de Amor Amazônia, Porto Velho, Rondônia
  - *X*CEPHO - Centro de Estudos e Pesquisas em Hematologia e Oncologia, Santo André, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo, São Paulo
- China (4):
  - Beijing Cancer Hospital, Beijing
  - West China Hospital - Sichuan University, Chengdu
  - Sun yat-sen University Cancer Center, Guangzhou
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
- Denmark (2):
  - Aarhus Universitetshospital, Aarhus N
  - Herlev Hospital, Herlev
- France (2):
  - Centre Leon Berard, Lyon
  - Gustave Roussy, Villejuif
- Germany (2):
  - Krankenhaus Martha-Maria Halle-Dölau, Klinik für Urologie, Halle
  - Martini-Klinik am UKE GmbH, Hamburg
- Greece (3):
  - Alexandras General Hospital of Athens, Athens
  - Attikon University General Hospital, Chaïdári
  - Theageneio Hospital, Thessaloniki
- Italy (8):
  - A.O. Universitaria Ospedale Consorziale Policlinico Di Bari, Bari, Apulia
  - Istituto Nazionale Tumori Irccs Fondazione G. Pascale, Napoli, Campania
  - Azienda Ospedaliero-Universitaria S.Orsola-Malpighi, Bologna, Emilia-Romagna
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola, Meldola, Emilia-Romagna
  - Policlinico Universitario "Agostino Gemelli", Rome, Lazio
  - Irccs Ospedale San Raffaele, Milan, Lombardy
  - Azienda Ospedaliera S. Maria - Terni, Terni, Umbria
  - IRCCS Istituto Oncologico Veneto (IOV), Padua, Veneto
- Health Pharma Professional Research, Mexico City, Mexico CITY (federal District), Mexico
- Poland (4):
  - Szpital Wojewódzki im. Miko?aja Kopernika, Koszalin
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Pratia Poznan, Późna
  - Szpital Grochowski im. dr med. Rafa?a Masztaka Sp. z o.o., Warsaw
- South Korea (6):
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (6):
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Institut Catala d Oncologia Hospital Duran i Reynals, Barcelona
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital de Madrid Norte Sanchinarro- Centro Integral Oncologico Clara Campal, Madrid
- Turkey (Türkiye) (5):
  - Adana Baskent University Medical Faculty, Adana
  - Ankara City Hospital, Ankara
  - Trakya Universitesi Tip Fakultesi, Medikal Onkoloji Bilim Dali, Balkan Yerleskesi, Edirne
  - Izmir Medical Point Hospital, Izmir
  - Goztepe Prof.Dr. Suleyman Yalcin City Hospital, Kadiköy
- United Kingdom (3):
  - Barts and the London NHS Trust, London
  - Royal Preston Hosptial, Preston
  - Royal Marsden Hospital (Sutton), Sutton

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing